CLINICAL TRIAL: NCT03369691
Title: Ethnic Influences on Stress, Energy Balance and Obesity in Adolescents
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Uma Rao, Professor, University of California, Irvine
Other Study IDs: 20173441
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Adolescent; Stress; Physical Activity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will examine the mechanisms linking race, stress and biobehavioral factors to energy balance and obesity in both natural and controlled environments in African-American and Caucasian adolescent females. A Hispanic/Latina cohort has recently been added with permission for the sponsor.

DETAILED DESCRIPTION:
Obesity is one of the most serious public health problems in the US; its prevalence has tripled in the last three decades and is associated with a range of short- and long-term medical and psychosocial problems. Adolescence is a critical period for the development and persistence of obesity, and is associated with changes in diet, physical activity and fitness, fat distribution and insulin sensitivity. There are racial and sex-specific disparities in the prevalence and burden of obesity. African-American (AA) females have the highest rates of obesity, and the clustered risk factors for coronary heart disease and metabolic syndrome are twice that of AA males. The reasons for racial and sex-specific disparities in the prevalence and burden of obesity are not well understood. AA experience higher stress levels than Non-Hispanic Whites (NHW) due to economic and social inequalities, and the effect of stress on energy-dense diet and adiposity is more prominent in females. A better understanding of the mechanisms that link stress to obesity, particularly during adolescence when high rates of obesity, increased stressful experiences and stronger behavioral and physiological responses to stress emerge, will contribute to new clinical guidelines for reducing obesity and associated medical conditions in AA females.

The Physiological stress system affects obesity and mediates its adaptive functions via hypothalamic-pituitary-adrenal (HPA) axis. Prolonged stress-induced glucocorticoid secretion promotes the consumption of energy-dense diet (EI) and abdominal fat deposition both directly and indirectly through its effects on metabolic hormones. Stress also reduces physical activity and alters energy balance. The proposed study will examine the effects of stress and HPA axis on EI and physical activity-related energy expenditure in 100 AA and 100 NHW adolescent females. The effects on EI will be assessed in two contexts, the natural environment and under controlled conditions incorporating a standardized psychosocial stressor. Stress will be assessed in the natural environment as multiple domains (i.e., individual, family and social), and several indices of the HPA axis will be obtained to represent diurnal variation, its status over 12-15 weeks and reactivity to stress. Obesity-related parameters will be measured through anthropometry, fat distribution and cardio-metabolic biomarkers.

Associations among stress, HPA activity/function, energy balance and obesity-related parameters will be compared between and within AA and NHW samples. In combination they will improve our understanding of the social factors and biobehavioral mechanisms of both racial and individual differences in obesity and facilitate the development of effective treatments within and across racial groups according to the principles of individualized medicine. To our knowledge, racial differences in objectively-measured diet intake and energy expenditure in response to stress, or their underlying physiological mechanisms, have not been assessed in adolescents or adults. This is an important knowledge gap in our efforts to develop better evidence-based translational obesity prevention and weight-control interventions as the traditional interventions are not effective with minority youth.

ELIGIBILITY:
Inclusion Criteria:

* African-American, Hispanic, Non-Hispanic White females from 13-17 years old and Tanner Stage ≥III.
* BMI values will be balanced (1/3rd normal, 1/3rd overweight and 1/3rd obese range percentile BMI values) using Center for Disease Control criteria

Exclusion Criteria:

* Participants with a BMI below the normal range, trying to lose weight, on medications that affect appetite or hypothalamic-pituitary-adrenal axis, or with a history of bariatric surgery, will be excluded.
* Restrained or binge eaters, individuals who score below 50 on a 100 mm Visual Analog Scale for foods provided in the study, or those allergic to these foods will be excluded.
* Participants with major psychiatric disorders (e.g., anxiety, eating, mood, substance use disorders) or medical problems (e.g., endocrine disorders or unstable cardiac, pulmonary or renal conditions) will be excluded.
* Pregnant females, or those suspected of being pregnant, will be excluded.

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Comparison of food intake from buffet lunch after the control and stress sessions | 7 days between the two sessions
  Randomize lab session to assign each participant to a non-stress or stress condition, and reversed in the next session. Ad-libitum food intake (amount of added sugar and solid fat) during both sessions will be measured and compared.

SECONDARY OUTCOMES:
Body mass index (BMI) | 1 hour
  Weight (kg) and height (inches) will be used to determine BMI in kg/cm^2
Physical activity energy expenditure | 7 days
  Average moderate and vigorous activity (minutes) will be recorded through the Actigraph device
Visceral fat percent | 1 hour
  Amount of visceral fat (percent of total fat) will be determined by dual-energy x-ray scan

CONTACTS AND LOCATIONS:
Overall Officials: Uma Rao, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Universty of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03369691/ICF_004.pdf